CLINICAL TRIAL: NCT01819922
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, Two-way Crossover Study To Assess The Effect Of Pf-05175157 As A Single Oral Dose On Metabolic And Cardiopulmonary Parameters During Steady State And Graded Exercise In Healthy Subjects
Brief Title: Effect Of Single-Dose PF-05175157 On Metabolic And Cardiopulmonary Parameters
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B1731008
Record Dates: First submitted 2013-02-24; First posted 2013-03-28 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Cardiopulmonary exercise testing; metabolic parameters; Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-05175157 (Experimental)
  Interventions: Drug: PF-05175157
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05175157 — 600 mg as powder in capsule, one dose within 5 minutes prior to AM meal
  Arms: PF-05175157
Drug: Placebo — Placebo powder in capsule, one dose within 5 minutes prior to AM meal
  Arms: Placebo

SUMMARY:
This study is designed to assess the effect of one single dose of PF-05175157 on metabolic and cardiopulmonary parameters before, during and after treadmill exercise in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non child bearing potential only, between the ages of 18 and 40 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 18 to 28 kg/m2; and a total body weight >50 kg (110 lbs).
* Subjects with maximum effort studies (peak RER >1.05) and normal exercise capacity as defined by peak VO2 ≥80% and ≤120% of predicted and no evidence of inducible ischemia or significant arrhythmia at the time of peak aerobic capacity testing 3 (±1) days prior to initiation of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* History of smoking in the past 5 years or history or evidence of habitual use of other (non smoked) tobacco or nicotine-containing products within 3 months of Screening or positive cotinine test at Screening or Day -3 (±1).
* Dry eye symptoms

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-05175157 Then Placebo: Participants who met the pre-defined cardiopulmonary exercise test (CPET) criteria, received single dose of PF-05175157 600 milligram (mg) capsule orally in first intervention period then single dose of placebo matched to PF-05175157 capsule, 600 mg orally in second intervention period. A washout period of at least 7-10 days was maintained between each intervention period.
- Placebo Then PF-05175157: Participants who met the pre-defined CPET criteria, received single dose of placebo matched to PF-05175157, 600 mg capsule orally in first intervention period then single dose of PF-05175157 600 mg capsule orally in second intervention period. A washout period at least of 7-10 days was maintained between each intervention period.
Period: First Intervention Period (1 Day)
Arm/Group | PF-05175157 Then Placebo | Placebo Then PF-05175157
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period (at Least 7-10 Days)
Arm/Group | PF-05175157 Then Placebo | Placebo Then PF-05175157
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention Period (1 Day)
Arm/Group | PF-05175157 Then Placebo | Placebo Then PF-05175157
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who performed the peak aerobic capacity test, were randomized and had at least 1 dose of randomized treatment.
Groups:
- Overall Participants: All randomized participants who received single dose of PF-05175157 600 mg capsule or single dose of placebo matched to PF-05175157 600 mg capsule in either first or second intervention period.
Arm/Group | Overall Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Oxygen Uptake Efficiency Slope (OUES) [Mean (Standard Deviation); unit: milliliter per log10*liter [mL/log10(L)]] | 3163.333 (3200.000)
Volume of oxygen [Mean (Standard Deviation); unit: milliliter per kilogram per minute] | 41.033 (3.6084)
Respiratory Exchange Ratio [Mean (Standard Deviation); unit: ratio] | 1.313 (0.0881)
Minute Ventilation and Carbon Dioxide Production (VE/VCO2 slope) [Mean (Standard Deviation); unit: unitless] | 20.800 (3.5545)
Volume of Oxygen (VO2) at Anaerobic Threshold [Mean (Standard Deviation); unit: milliliter (mL)] | 19.467 (2.6800)
Oxygen pulse [Mean (Standard Deviation); unit: milliliter per beat (mL/beat)] | 16.808 (2.0518)
Aerobic Efficiency [Mean (Standard Deviation); unit: milliliter per watt (mL/watt)] | 10.442 (0.8544)
Physical Work Capacity [Mean (Standard Deviation); unit: beats per minute (bpm)] | 154.750 (25.3094)

OUTCOME MEASURES:

1. Primary Outcome: Systolic Function: Global Longitudinal Left Ventricular (LV) Strain: 20 Minutes Pre-dose
Description: Global longitudinal left ventricular strain was defined as the percent change in left ventricular longitudinal dimension in comparison to its original dimension. Global longitudinal LV strain was assessed by echocardiography using speckled tracking analysis.
Time Frame: 20 minutes pre-dose
Population: Full analysis set (FAS) was defined as all participants who performed the peak aerobic capacity test, were randomized and received at least 1 dose of randomized treatment, and had at least 1 pharmacodynamic (PD) measurement.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- PF-05175157 600 mg: Participants who met the pre-defined CPET criteria received single dose of PF-05175157 600 mg capsule orally in either first or second intervention period. A washout period of at least 7-10 days was maintained between each intervention period.
- Placebo: Participants who met the pre-defined CPET criteria received single dose of placebo matched to PF-05175157 600 mg capsule orally in either first or second intervention period. A washout period of at least 7-10 days was maintained between each intervention period.
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
percent change | -19.779 (1.9682) | -20.483 (2.0050)

2. Primary Outcome: Systolic Function: Global Longitudinal Left Ventricular (LV) Strain: 1 Hour 30 Minutes Post-dose
Description: as for outcome 1
Time Frame: 1 hour 30 minutes post-dose
Population: FAS was defined as all participants who performed the peak aerobic capacity test, were randomized and received at least 1 dose of randomized treatment, and had at least 1 PD measurement.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
percent change | -19.728 (2.0187) | -20.183 (2.0058)

3. Primary Outcome: Systolic Function: Global Longitudinal Left Ventricular (LV) Strain: 2 Hours 5 Minutes Post-dose
Description: as for outcome 1
Time Frame: 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
percent change | -24.058 (2.9330) | -24.587 (3.5740)

4. Primary Outcome: Cardiopulmonary Exercise Test: Oxygen Uptake Efficiency Slope (OUES): 1 Hour 40 Minute Post-dose
Description: OUES was defined as an index of cardiopulmonary functional reserve that was based upon a submaximal exercise effort. OUES relates oxygen uptake to total ventilation during exercise.
Time Frame: 1 hour 40 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/log10(L)
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
mL/log10(L) | 3192.500 (458.6170) | 3165.833 (439.0373)

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event. Treatment-emergent were events between first dose of study drug and up to 5-10 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. Adverse events included both serious and non-serious adverse events.
Time Frame: Baseline up to 5-10 days after last dose of study drug (up to 25 days)
Population: Safety analysis set was defined as all participants who performed the peak aerobic capacity test, were randomized and who had received at least 1 dose of randomized treatment.
Measure: Number; unit: participants
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
participants
  Adverse events | 0 | 2
  Serious adverse events | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Criteria for clinically significant:Hematology (hemoglobin,hematocrit,red blood corpuscles [RBC] count:less than [<]0.8*lower limit of normal [LLN];platelets:<0.5*LLN/greater than [>]1.75*upper limit of normal [ULN];white blood corpuscles [WBC]:<0.6*LLN or >1.5*ULN;lymphocytes, total neutrophils:<0.8*LLN or >1.2*ULN;basophils,eosinophil, monocytes:>1.2*ULN);Liver Function(aspartate aminotransferase, alanine aminotransferase,alkaline phosphatase:>0.3*ULN;total protein,albumin:<0.8*LLN or >1.2*ULN;total bilirubin:>1.5*ULN);Renal Function (blood urea nitrogen,creatinine:>1.3*ULN; uric acid:>1.2*ULN);Electrolytes (sodium:<0.95*LLN or >1.05*ULN,potassium,chloride, calcium,bicarbonate:<0.9*LLN or >1.1*ULN; glucose fasting:<0.6*LLN or >1.5*ULN);Urinalysis (urine pH:>1.5*ULN or >4.5;urine glucose,ketones,proteins, nitrites, leukocyte esterase,blood/hemoglobin:greater than or equal to (>=)1;urine WBC and RBC,urine bacteria:>=20/High Power Field [HPF];epithelial cells:>=6/HPF).
Time Frame: Baseline up-to 3 hours post-dose
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
participants | 4 | 6

7. Secondary Outcome: Number of Participants With Categorical Post-dose Cardiovascular Monitoring Data
Description: Participants who met the pre-defined criteria for clinically significant cardiovascular events were reported. Criteria for clinically significant cardiovascular events: Blood pressure (BP) [supine systolic and sitting systolic BP (SBP): <90 millimeter of mercury (mm Hg), >=30 mmHg maximum increase and decrease from baseline in same posture; supine diastolic and sitting diastolic BP (DBP): <50 mm Hg, >=20 mmHg maximum increase and >=30 mmHg maximum decrease from baseline in same posture]; pulse rate: supine and sitting: <40 or >120 bpm.
Time Frame: Baseline up-to 3 hours post-dose
Population: Safety analysis set was defined as all participants who performed the peak aerobic capacity test, were randomized and who had received at least 1 dose of randomized treatment. Here, "n" specified the number of participants who were evaluable for the specified criteria.
Measure: Number; unit: participants
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
participants
  Supine SBP (n=12) | 0 | 0
  Supine DBP (n=12) | 0 | 0
  Supine pulse rate (n=12) | 0 | 0
  Sitting pulse rate (n=1) | 0 | 0
  Sitting SBP (n=1) | 0 | 0
  Sitting DBP (n=1) | 0 | 0
  Supine SBP: Maximum Increase from Baseline (n=12) | 0 | 0
  Supine DBP: Maximum increase from baseline (n=12) | 0 | 1
  Supine SBP: Maximum decrease from baseline (n=12) | 0 | 0
  Supine DBP: Maximum decrease from baseline (n=12) | 0 | 0

8. Secondary Outcome: Number of Participants With Categorical Post-dose Cardiovascular Monitoring Data: Electrocardiogram (ECG) Parameters
Description: Criteria for clinically significant ECG values included: maximum PR interval >=300 millisecond (msec) and maximum increase of >=25 percent (%) from baseline value of >200 msec and >=50 % for baseline value of <=200 msec, maximum QRS interval >=140 msec or maximum increase of >=50% for baseline value of >100 msec; QT interval corrected using the Fridericia formula (QTcF) 450-<480 msec, 480-<500, >=500 msec or increase of >45 msec or maximum increase of >=30 to <60 and >=60 msec for QT interval where, PR interval: interval between the start of the P wave and the start of the QRS complex corresponding to the time between the onset of atrial depolarization and onset of ventricular depolarization; QRS interval: time from electrocardiogram Q wave to the end of the T wave corresponding to ventricle depolarization, QTcF interval: time corresponding to the beginning of depolarization to repolarization of the ventricles.
Time Frame: Baseline up-to 3 hour post-dose
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
participants
  Maximum PR interval >=300 msec | 0 | 0
  Maximum QRS complex >=140 msec | 0 | 0
  Maximum QTCF interval 450-<480 msec | 1 | 0
  Maximum QTCF interval 480-<500 msec | 0 | 0
  Maximum QTCF interval >=500 msec | 0 | 1
  PR interval increase from baseline >=25/50% | 0 | 0
  QRS complex increase from baseline >=50% | 0 | 0
  QTCF interval increase from baseline>=30 to<60msec | 0 | 3
  QTCF interval increase from baseline >=60 msec | 1 | 1

9. Secondary Outcome: Cardiopulmonary Exercise Test: Peak Volume of Oxygen (VO2)
Description: VO2 was the maximum rate of oxygen consumption as measured during incremental or prolonged, sub-maximal exercise. It reflects the aerobic physical fitness of the individual. It was assessed during indirect measure of heat production (calorimetry). The unit of measure is milliliter per kilogram per minute (mL/kg/min).
Time Frame: 1 hour 40 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
mL/kg/min | 41.325 (3.9857) | 42.092 (4.4663)

10. Secondary Outcome: Cardiopulmonary Exercise Test: Respiratory Exchange Ratio (RER)
Description: RER was defined as the ratio between the amount of oxygen (O2) consumed and carbon dioxide (CO2) produced in one breath. The parameter was assessed during indirect measure of heat production (calorimetry).
Time Frame: 1 hour 40 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
ratio | 0.984 (0.1289) | 1.013 (0.1462)

11. Secondary Outcome: Cardiopulmonary Exercise Test: Minute Ventilation and Carbon Dioxide Production (VE/VCO2 Slope)
Description: VE/VCO2 slope was also termed as ventilator efficiency. It was defined as the amount of minute ventilation required to eliminate 1 liter of carbon dioxide. The determinants of VE/VCO2 included fractional dead space and partial pressure of carbon dioxide. The parameter was assessed during indirect calorimetry.
Time Frame: 1 hour 40 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
unitless | 22.325 (4.0815) | 21.375 (3.3759)

12. Secondary Outcome: Cardiopulmonary Exercise Test: Volume of Oxygen (VO2) at Anaerobic Threshold (AT)
Description: VO2 at anaerobic threshold was widely recognized as a sub-max indicator of fitness. The parameter was assessed during indirect calorimetry.
Time Frame: 1 hour 40 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
mL | 19.008 (3.5279) | 18.633 (4.0130)

13. Secondary Outcome: Cardiopulmonary Exercise Test: Oxygen (O2) Pulse
Description: Oxygen Pulse (VO2 /Heart Rate) was equal to stroke volume multiplied by oxygen extraction. This parameter was assessed during cardiopulmonary exercise test.
Time Frame: 1 hour 40 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
mL/beat | 16.692 (2.2342) | 16.850 (2.3781)

14. Secondary Outcome: Cardiopulmonary Exercise Test: Oxygen (O2) Kinetics
Description: Oxygen kinetics describes the dependence of respiration of isolated cells on oxygen partial pressure. The characteristics of oxygen uptake kinetics differ with intensity of exercise.
Time Frame: 1 hour 40 minutes post-dose
Population: Data was not collected for this outcome measure as per study team's decision since single dose was not considered to be sufficient to analyze this specific parameter.
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Cardiopulmonary Exercise Test: Aerobic Efficiency
Description: Aerobic efficiency was defined as volume of oxygen divided by work. This parameter was assessed during cardiovascular exercise test.
Time Frame: 1 hour 40 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/watt
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
mL/watt | 10.358 (0.6201) | 10.483 (0.7638)

16. Secondary Outcome: Cardiopulmonary Exercise Test: Physical Work Capacity at a Heart Rate of 130 Beats Per Minute (PWC 130)
Description: Physical work capacity evaluates the capacity of an individual to perform physically demanding work tasks. PWC 130 was a simple sub-max exercise parameter that can be used as surrogate for fitness that was independent of metabolic cart measurements. Interventions that improve fitness improve the PWC 130.
Time Frame: 1 hour 40 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
bpm | 156.583 (31.4078) | 156.667 (26.7185)

17. Secondary Outcome: Cardiac Structure: Left Ventricular Volume
Description: Left ventricular volume was defined as volume of blood pumped from the left ventricle to the heart per beat. It was calculated using measurements of ventricle volumes from an echocardiogram and subtracting the volume of the blood in the ventricle at the end of a beat (called end-systolic volume) from the volume of blood just prior to the beat (called end-diastolic volume). Left ventricular volume was reported using modified Simpson's technique.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
mL
  20 minutes pre-dose | 76.750 (10.9555) | 76.333 (11.8117)
  1 hour 30 minutes post-dose | 77.167 (12.2610) | 77.333 (11.9494)
  2 hours 5 minutes post-dose | 85.250 (15.2442) | 85.000 (13.6980)

18. Secondary Outcome: Change From Baseline in the Left Ventricular Volume
Description: Left ventricular volume was defined as volume of blood pumped from the left ventricle to the heart per beat. It was calculated using measurements of ventricle volumes from an echocardiogram and subtracting the volume of the blood in the ventricle at the end of a beat (called end-systolic volume) from the volume of blood just prior to the beat (called end-diastolic volume). Change from baseline in left ventricular volume was reported using modified Simpson's technique.
Time Frame: 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
mL
  Change at 1 hour 30 minutes post-dose | 0.417 (3.6546) | 1.000 (3.1909)
  Change at 2 hours 5 minutes post-dose | 8.500 (8.5546) | 8.667 (8.0265)

19. Secondary Outcome: Cardiac Structure: Left Ventricular Wall Thickness
Description: Left ventricle is the chamber in the heart responsible for pumping blood to the rest of the body. Thickening of the lower chambers of left ventricular wall is also termed as ventricular hypertrophy. It was assessed by echocardiography using 2-dimensional gray-scale imaging; M-mode.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 14
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Cardiac Structure: Left Ventricular Geometry
Description: Left ventricular geometry was assessed by echocardiography using 2-dimensional gray-scale imaging. Relative wall thickness was the index of left ventricular geometry and defined as the sum of interventricular septal thickness (mm) and posterior wall thickness (mm) divided by LV internal end-diastolic diameter (mm).
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 14
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Cardiac Structure: Right Ventricular Dimension
Description: Right ventricle is the chamber in the heart responsible for pumping blood to the lungs. Right ventricular dimensions included end-diastole area (EDA) and end-systole area (ESA). It was assessed by echocardiography using 2-dimensional gray-scale imaging.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimetre (mm)
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
millimetre (mm)
  End-diastole area: 20 minutes pre-dose | 24.250 (2.4693) | 23.704 (2.8601)
  End-diastole area: 1 hour 30 minutes post-dose | 24.408 (2.4247) | 23.975 (2.7877)
  End-diastole area: 2 hours 5 minutes post-dose | 24.203 (2.0097) | 23.642 (2.1318)
  End-systole area: 20 minutes pre-dose | 14.675 (2.4643) | 13.992 (2.3971)
  End-systole area: 1 hour 30 minutes post-dose | 14.350 (2.2841) | 14.342 (2.1923)
  End-systole area: 2 hours 5 minutes post-dose | 10.783 (2.0395) | 10.208 (1.8569)

22. Secondary Outcome: Change From Baseline in Right Ventricular Dimension
Description: Right ventricle is the chamber in the heart responsible for pumping blood to the lungs. Right ventricular dimensions included end-diastole area and end-systole area. It was assessed by echocardiography using 2-dimensional gray-scale imaging. Change from baseline in right ventricular dimension was reported.
Time Frame: 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
mm
  EDA: change at 1hour 30 minutes post-dose | 0.158 (0.8350) | 0.271 (1.0015)
  EDA: change at 2 hours 5 minutes post-dose | -0.047 (1.2544) | -0.062 (2.1118)
  ESA: change at 1 hour 30 minutes post-dose | -0.325 (0.7533) | 0.350 (0.4622)
  ESA: change at 2 hours 5 minutes post-dose | -3.892 (1.9351) | -3.783 (1.7497)

23. Secondary Outcome: Cardiac Structure: Atrial Volume
Description: Atrial volumes were assessed by echocardiography using 2-dimensional gray-scale imaging and were calculated using the bi-plane area-length method. Both end-systole volumes (ESV) and end-diastole volumes (EDV) were reported.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
mL
  End-diastole: 20 minutes pre-dose | 47.000 (12.7422) | 50.750 (10.4544)
  End-diastole:1 hour 30 minutes post-dose | 47.000 (11.2896) | 49.833 (10.0890)
  End-diastole: 2 hours 5 minutes post-dose | 42.917 (9.9312) | 44.917 (9.7650)
  End-systole: 20 minutes pre-dose post-dose | 19.917 (6.7347) | 20.083 (4.8328)
  End-systole:1 hour 30 minutes post-dose | 21.333 (6.8667) | 21.417 (4.6993)
  End-systole: 2 hours 5 minutes post-dose | 16.417 (5.6642) | 16.083 (3.3428)

24. Secondary Outcome: Change From Baseline in Atrial Volumes
Description: Atrial volumes were assessed by echocardiography using 2-dimensional gray-scale imaging and were calculated using the bi-plane area-length method. Both end-systole volumes and end-diastole volumes were reported. Change from baseline in atrial volume was reported.
Time Frame: 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
mL
  EDV: change at 1 hour 30 minute post-dose | 0.000 (2.7303) | -0.917 (1.6214)
  EDV: change at 2 hours 5 minute post-dose | -4.083 (4.7950) | -5.833 (5.2886)
  ESV: change at 1 hour 30 minute post-dose | 1.417 (1.8809) | 1.333 (1.5570)
  ESV: change at 2 hours 5 minutes post-dose | -3.500 (2.3160) | -4.000 (3.9312)

25. Secondary Outcome: Systolic Function: Ejection Fraction
Description: Systolic ejection fraction was the fraction of the end-diastolic volume (EDV) that was ejected out of left ventricle with each contraction, estimated by echocardiography. EDV was the volume of blood within a ventricle immediately before a contraction. Ejection fraction served as a general measure of the cardiac function of a participant.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of EDV
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
percentage of EDV
  20 minutes pre-dose | 63.190 (5.9675) | 63.058 (6.3917)
  1 hour 30 minutes post-dose | 62.525 (5.6452) | 62.633 (6.5173)
  2 hours 5 minutes post-dose | 72.462 (5.8507) | 72.949 (5.1819)

26. Secondary Outcome: Change From Baseline in Ejection Fraction
Description: Systolic ejection fraction was the fraction of the end-diastolic volume that was ejected out of left ventricle with each contraction, estimated by echocardiography. EDV was the volume of blood within a ventricle immediately before a contraction. Ejection fraction served as a general measure of the cardiac function of a participant. Change from baseline in ejection fraction was reported.
Time Frame: 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of EDV
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
percentage of EDV
  Change at 1 hour 30 minutes post-dose | -0.665 (2.3178) | -0.426 (1.7638)
  Change at 2 hours 5 minutes post-dose | 9.272 (5.0915) | 9.891 (5.6629)

27. Secondary Outcome: Systolic Function: Peak Contractile Velocity
Description: It was assessed by echocardiography using Tissue Doppler Imaging (Color Post-Processing).
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeter per second (cm/sec)
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
centimeter per second (cm/sec)
  20 minutes pre-dose | 7.625 (1.0997) | 9.025 (2.0521)
  1 hour 30 minutes post-dose | 7.758 (1.4457) | 9.083 (1.8075)
  2 hours 5 minutes post-dose | 12.875 (1.4085) | 13.925 (1.3903)

28. Secondary Outcome: Change From Baseline in Peak Contractile Velocity
Description: It was assessed by echocardiography using Tissue Doppler Imaging (Color Post-Processing). Change from baseline in peak contractile velocity was reported.
Time Frame: 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
cm/sec
  Change at 1 hour 30 minutes post-dose | 0.133 (0.6541) | 0.058 (0.4295)
  Change at 2 hours 5 minutes post-dose | 5.250 (1.6963) | 4.900 (2.0476)

29. Secondary Outcome: Systolic Function: Rotation/Torsion
Description: Torsion is the twisting of an object due to an applied torque. It is expressed in newton metres. The left ventricle twists in systole storing potential energy and untwists (recoils) in diastole releasing the energy. Twist aids left ventricular ejection and untwist aids relaxation and ventricular filling. Therefore, rotation and torsion are important in cardiac mechanics. It was assessed by echocardiography using speckled tracking analysis .
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 14
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Systolic Function: Global Strain Rate
Description: Global longitudinal left ventricular strain rate was defined as the rate of percent change in left ventricular longitudinal dimension in comparison to its original dimension. Global strain rate was assessed by echocardiography using speckled tracking analysis.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change per second
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
percent change per second
  20 minutes pre-dose | -1.043 (0.1449) | -1.124 (0.1756)
  1 hour 30 minutes post-dose | -1.047 (0.1462) | -1.078 (0.1171)
  2 hours 5 minutes post-dose | -1.845 (0.5499) | -1.916 (0.5786)

31. Secondary Outcome: Change From Baseline in Systolic Global Strain Rate
Description: Global longitudinal left ventricular strain rate was defined as the rate of percent change in left ventricular longitudinal dimension in comparison to its original dimension. Global strain rate was assessed by echocardiography using speckled tracking analysis. Change from baseline in systolic global strain rate was reported.
Time Frame: 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change per second
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
percent change per second
  Change at 1 hour 30 minutes post-dose | -0.003 (0.1208) | 0.047 (0.1070)
  Change at 2 hours 5 minutes post-dose | -0.802 (0.5884) | -0.792 (0.5934)

32. Secondary Outcome: Trans-mitral Doppler: Ratio
Description: Trans-mitral doppler ratio was Transmitral E wave peak velocity divided by transmitral A wave peak velocity. The E/A ratio was defined the ratio of the early (E) to late (A) ventricular filling velocities and was marker of the function of the left ventricle of the heart. It was determined on spectral doppler echocardiography.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes
Population: FAS was defined as all participants who performed the peak aerobic capacity test, were randomized and received at least 1 dose of randomized treatment, and had at least 1 PD measurement. Here, "n" specified the number of participants who were evaluable for the specified time-point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
ratio
  20 minutes pre-dose (n=12, 12) | 186.894 (53.0097) | 182.236 (39.8589)
  1 hour 30 minutes post-dose (n=12, 12) | 184.050 (40.4499) | 190.424 (36.1174)
  2 hours 5 minutes post-dose (n=11, 11) | 134.205 (52.0345) | 125.156 (34.6253)

33. Secondary Outcome: Change From Baseline in Trans-mitral Doppler Ratio
Description: Trans-mitral doppler ratio was Transmitral E wave peak velocity divided by transmitral A wave peak velocity. The E/A ratio was defined the ratio of the early (E) to late (A) ventricular filling velocities and was marker of the function of the left ventricle of the heart. It was determined on spectral doppler echocardiography. Change from baseline in trans-mitral ration was reported.
Time Frame: 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
ratio
  Change at 1 hour 30 minutes post-dose (n=12,12) | -2.844 (17.6282) | 8.188 (19.7236)
  Change at 2 hours 5 minutes post-dose (n=11,11) | -57.803 (62.4623) | -61.330 (44.7622)

34. Secondary Outcome: Trans-mitral Doppler: Time
Description: Trans-mitral doppler time was measured as the time between the closure of the aortic valve and the opening of the mitral valve. It was determined on spectral doppler echocardiography.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
msec
  20 minutes pre-dose (n=12, 12) | 168.333 (24.6810) | 158.917 (19.8470)
  1 hour 30 minutes post-dose (n=12, 12) | 166.417 (19.0333) | 160.750 (16.8799)
  2 hours 5 minutes post-dose (n=11, 11) | 179.091 (25.8204) | 173.727 (30.7542)

35. Secondary Outcome: Change From Baseline in Trans-mitral Doppler Time
Description: Trans-mitral doppler time was measured as the time between the closure of the aortic valve and the opening of the mitral valve. It was determined on spectral doppler echocardiography. Change from baseline in trans-mitral doppler time was reported.
Time Frame: 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
msec
  Change at 1 hour 30 minutes post-dose (n=12, 12) | -1.917 (8.2513) | 1.833 (6.1472)
  Change at 2 hours 5 minutes post-dose (n=11, 11) | 11.273 (29.3465) | 14.273 (44.1001)

36. Secondary Outcome: Early and Late Peak Tissue Velocity
Description: Tissue velocities were measured off-line from two dimensional (2D) color-coded tissue doppler images and reported as the average of 3 consecutive cardiac cycles. Tissue Doppler Imaging measured the velocity of the heart muscle or myocardium through the phases of one or more heartbeats by the Doppler effect (frequency shift) of the reflected ultrasound. Early and late peak tissue velocities (EPV and LPV) were reported.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
cm/sec
  EPV: 20 minutes pre-dose (n=12, 12) | 9.892 (0.6934) | 10.375 (1.1663)
  EPV: 1 hour 30 minutes post-dose (n=12,12) | 10.017 (0.6939) | 10.342 (1.2132)
  EPV: 2 hours 5 minutes post-dose (n=12,12) | 11.600 (1.4635) | 11.825 (1.7889)
  LPV: 20 minutes pre-dose (n=12,12) | 5.233 (1.0210) | 5.375 (0.5754)
  LPV: 1 hour 30 minutes post-dose(n=12,12) | 4.933 (1.1555) | 5.500 (0.7058)
  LPV: 2 hours 5 minutes post-dose (n=8,9) | 6.688 (2.2599) | 6.544 (1.4800)

37. Secondary Outcome: Change From Baseline in Early and Late Peak Velocity
Description: Tissue velocities were measured off-line from 2D color-coded tissue doppler images and reported as the average of 3 consecutive cardiac cycles. Tissue Doppler Imaging measured the velocity of the heart muscle or myocardium through the phases of one or more heartbeats by the Doppler effect (frequency shift) of the reflected ultrasound. Change from baseline in early and late peak tissue velocities were reported.
Time Frame: 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 12 | 12
cm/sec
  EPV:change at1 hour 30 minutes post-dose(n=12,12) | -0.300 (0.4045) | 0.125 (0.4288)
  EPV:change at 2 hours 5 minutes post-dose(n= 8,9) | 1.713 (1.7008) | 1.144 (1.1780)
  LPV:change at1 hour 30 minute post-dose(n= 12,12) | 0.125 (0.3494) | -0.033 (0.2640)
  LPV:change at 2 hours 5 minutes post-dose(n=12,12) | 1.708 (1.1611) | 1.450 (1.1213)

38. Secondary Outcome: Diastolic Strain Rate
Description: Diastolic strain rate was defined as the rate of percent change in all segments of left ventricular dimension in comparison to its original dimension. It was assessed by echocardiography using speckled tracking analysis.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 14
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Peak Diastolic Untwisting Rate
Description: Diastolic untwisting is an important component of early diastolic left ventricular filling. Left ventricular diastolic function is determined by early diastolic relaxation and myocardial stiffness. Peak diastolic untwisting rate is defined as the rate of left ventricular relaxation. It was assessed by echocardiography using speckled tracking analysis.
Time Frame: 20 minutes pre-dose, 1 hour 30 minutes and 2 hours 5 minutes post-dose
Population: as for outcome 14
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Plasma Metabolomic Profiles Before and Immediately Following Steady State and Incremental Exercise
Description: Plasma metabolomic profiles before and immediately following steady state and incremental exercise were collected using vacutainer tube containing dipotassium ethylenediamine tetraacetic Acid (K2EDTA) were processed by the clinical site according to handling specifications.
Time Frame: 1 hour pre-dose, 1 hour 20 minutes and 2 hours 10 minutes post-dose
Population: as for outcome 14
Arm/Group | PF-05175157 600 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | PF-05175157 600 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05175157 600 mg (N=12) | Placebo (N=12)
Dizziness (Nervous system disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.